CLINICAL TRIAL: NCT02294084
Title: The Effect of Sitagliptin on Brown Adipose Tissue and Whole-body Metabolism in Overweight Pre-diabetic Men
Brief Title: Sitagliptin and Brown Adipose Tissue
Acronym: Sita01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ingrid Jazet (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Ingrid Jazet, Dr, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P14.242
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Neoplasms, Adipose Tissue
MeSH Terms: conditions — Neoplasms, Adipose Tissue | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Subjects will receive Sitagliptin in a dosage of 100 mg/day p.o. for 12 weeks. The dosage corresponds to 1 gift/day.
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Subjects will receive placebo for 12 weeks. Placebo will be given in 1 gift/day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sitagliptin — Each subject in this arm will receive Sitagliptin (100mg/day) for a duration of 12 weeks.
  Other Names: Januvia
  Arms: Sitagliptin
Drug: placebo — Each subject will receive a placebo (once a day) for 12 weeks.
  Arms: Placebo

SUMMARY:
The obesity epidemic has resulted in an exponential increase in obesity-related disorders including type 2 diabetes, dyslipidemia and cardiovascular disease. The associated morbidity and mortality have major consequences both at an individual as well as on the socioeconomical level. Thus, the development of novel therapies aimed at reducing the development of obesity is highly warranted. Brown adipose tissue (BAT) recently emerged as a novel player in energy expenditure in humans as it combusts fatty acids towards heat. Interestingly, obese subjects have less BAT as compared to lean subjects and activation of BAT by means of intermittent cold exposure reduces fat mass. Therefore, BAT is considered a promising novel target to reduce obesity and associated disorders. As cold exposure is not the most desired therapeutic strategy for humans, current pre-clinical research focuses on pharmacological activation of BAT.

Interestingly, the investigators have recently shown that central agonism of the receptor for the incretin hormone glucacon-like peptide-1 (GLP-1) results in activation of BAT in mice. One of the currently used anti-diabetic drugs that enhances GLP-1 availability is Sitagliptin (STG). Interestingly, STG also reduces body weight and plasma triglyceride (TG) levels in type 2 diabetes mellitus (T2DM) patients. The mechanism underlying these beneficial metabolic effects is currently unknown. The investigators hypothesize that STG enhances BAT activation, thereby increasing energy expenditure and combustion of TG-derived fatty acids, resulting in lowering of plasma TG levels and body weight.

To this end, the investigators will perform a randomized double-blinded placebo-controlled study in which 30 male Dutch Caucasian adults aged 35-50 years with moderate obesity and pre-diabetes are included. Subjects will be treated for 12 weeks with STG or placebo. Before and after treatment, the investigators will determine BAT volume and total BAT activity via cold-induced 18F-FDG PET-CT scans, resting energy expenditure via indirect calorimetry using ventilated hoods, body weight, and body composition via DEXA scan. Furthermore, before and after treatment, blood samples will be taken to measure plasma lipids, glucose and insulin levels.

This study will offer valuable novel insight in the effects of pharmacological activation of BAT in human obese subjects.

DETAILED DESCRIPTION:
In the current study, the effect of 12 weeks of STG treatment (100 mg/day p.o.) versus placebo will be studied in moderately obese pre-diabetic Dutch Caucasians males (35-50 years).

All study subjects will be screened and if the subject meets all the inclusion criteria, is willing to participate in the study and has signed the informed consent, he will be included. All subjects will be asked not to make any changes in their usual diets and physical activities before the start of the whole study. Subjects will undergo two study days (day 1 and day 2) before STG or placebo treatment and two study days after treatment (day 84 and day 85) on which a cold-induced PET-CT scan as well as metabolic studies and skeletal muscle biopsies are performed.

At screening a thorough medical history (see Appendix D) and physical examination will be performed. Subjects will be examined while in the fasting state. Anthropometric measurements will be performed as well as a basal blood sample will be taken by means of a venapunction. Basal blood measurements include hematology and kidney, liver, thyroid and lipid parameters as well as glucose, C-peptide and insulin concentrations. Thereafter, subjects ingest 75 grams of glucose orally (t=0) and at t=120 minutes a blood sample for the determination of glucose, C-peptide and insulin will be drawn (venapunction) to assess glucose tolerance.

On study days 1 and 84, which take place at the dept. of Nuclear Medicine in the Rijnland hospital, anthropometric measurements will be performed first, followed by ingestion of a CoreTemp Pill for core temperature registration application, a DEXA scan, and application of wireless iButtons to monitor skin temperature. Next, subjects will lay in a bed between two water-perfused matrasses and water temperature will be set at 32°C (= thermoneutrality). After 30 min of thermoneutrality, resting energy expenditure (REE) will be measured via ventilated hoods. Then, thermoneutral venous blood samples will be obtained. Water temperature will be gradually decreased and stabilized just above shivering level to induce maximum non-shivering thermogenesis (NST) for the next two hours. During the cooling period, blood pressure, heart rate and shivering are monitored at fixed intervals. At t=60 min, after one hour of stable cooling, 110 MBq (2.09 mSv) 18F-fluorodeoxyglucose (FDG) will be injected. At t=90 min, REE will be measured again. At t=120 min, cold-induced venous blood samples will be obtained followed by performance of the PET-CT scan (see Appendix B for an overview of study days 1 and 84).

On study days 2 and 85, which will be performed at the research laboratory at the LUMC, a muscle biopsy will be taken first. Then, after 1 hour of rest, an OGTT will be performed. To this end, a glucose drink containing 75 g of glucose will be ingested in maximum 5 minutes and at t=-10, 0, 10, 20, 30, 40, 50, 60, 90 and 120 min venous samples will be taken to assess glucose, insulin and C-peptide levels (see Appendix C for an overview of study days 2 and 85).

During the treatment period, study subjects will be called weekly by the researcher to ask for possible side effects, signs of hypoglycemia, plasma glucose levels (via finger prick, which will be done by the study subject himself) and compliance. Once a month, the study subject will return to the research laboratory at the LUMC. During this occasion, next to the above-mentioned parameters, also a venous blood sample will be obtained (venapunction) to assess plasma glucose, insulin and triglyceride levels.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers, Caucasians, born in the Netherlands
* Age: 35-55 years
* BMI > 25 and < 32 kg/m2
* plasma glucose levels 2 h after OGTT between 7.8 and 11 mM (e.g. impaired glucose tolerance)

Exclusion Criteria:

* Diabetes mellitus (determined on basis of oral glucose tolerance test (OGTT)) defined by ADA criteria
* BMI > 30 kg/m2 or < 25 kg/m2
* plasma glucose levels 2 h after OGTT < 7.8 or > 11.1 mM
* use of medication known to influence glucose and/or lipid metabolism or BAT activity (e.g. beta blockers)
* any significant chronic disease
* renal, hepatic or endocrine disease
* smoking
* participation in an intensive weight-loss program or vigorous exercise program during the last year before start of the study
* difficulties to insert an intravenous catheter
* recent participation in other research projects (within the last 3 months)

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The effect of sitagliptin treatment on BAT activity in overweight, pre-diabetic subjects BAT volume and activity will be measured by means of cold-induced 18F-FDG PET-CT scans | after 12 weeks of treatment
  BAT volume and activity will be measured by means of cold-induced 18F-FDG PET-CT scans

SECONDARY OUTCOMES:
The effect of sitagliptin treatment on energy expenditure in overweight, pre-diabetic subjects indirect calorimetrie | after 12 weeks of treatment
  indirect calorimetrie
The effect of sitagliptin treatment on muscle glucose metabolism in overweight, pre-diabetic subjects Expression and/or activation of biomarkers for insulin signaling and glucose and lipid metabolism in skeletal muscle biopsies | after 12 weeks of treatment
  Expression and/or activation of biomarkers for insulin signaling and glucose and lipid metabolism in skeletal muscle biopsies
The effect of sitagliptin treatment on fat mass in overweight, pre-diabetic subjects Fat mass will be measured via DEXA scan | after 12 weeks of treatment
  Fat mass will be measured via DEXA scan
The effect of sitagliptin treatment on glucose metabolism in overweight, pre-diabetic subjects serum glucose, insulin, and HbA1c. Furthermore, insulin secretion will be determined by OGTT together with C-peptine, glucose and insulin area under the curve | after 12 weeks of treatment
  We will assess fasting serum glucose, insulin, and HbA1c. Furthermore, insulin secretion will be determined by OGTT together with C-peptine, glucose and insulin area under the curve
The effect of sitagliptin treatment on plasma lipid levels in overweight, pre-diabetic subjects total cholesterol, HDL-C LDL-C triglycerides, and free fatty acids in plasma | after 12 weeks of treatment
  We will assess total cholesterol, HDL-C LDL-C triglycerides, and free fatty acids in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Rensen, PhD, Principal Investigator — Head of department
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nahon KJ, Doornink F, Straat ME, Botani K, Martinez-Tellez B, Abreu-Vieira G, van Klinken JB, Voortman GJ, Friesema ECH, Ruiz JR, van Velden FHP, de Geus-Oei LF, Smit F, Pereira Arias-Bouda LM, Berbee JFP, Jazet IM, Boon MR, Rensen PCN. Effect of sitagliptin on energy metabolism and brown adipose tissue in overweight individuals with prediabetes: a randomised placebo-controlled trial. Diabetologia. 2018 Nov;61(11):2386-2397. doi: 10.1007/s00125-018-4716-x. Epub 2018 Aug 25. PMID 30145664
- Available data/document: Clinical Study Report — https://www.health-holland.com/project/2015/effect-of-antidiabetic-drug-on-brown-adipose-tissue-bat-in-overweight-men — A simplified summary of the main results of the study can be found when following the link. In addition, the results are described in a paper that will be published by Diabetologia later this year.